CLINICAL TRIAL: NCT01239212
Title: Pharmacokinetics and Safety of 50 mg/kg IV Levetiracetam (Keppra) in Full Term and Preterm Neonates
Brief Title: Dosing of Levetiracetam (Keppra) in Neonates
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Stephanie Merhar, MD, Assistant Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101335
Record Dates: First submitted 2010-10-28; First posted 2010-11-11 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Seizures
Keywords: seizures; neonate; levetiracetam; Epilepsy; central nervous system diseases; anticonvulsants
MeSH Terms: conditions — Seizures; Epilepsy; Central Nervous System Diseases | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: levetiracetam — 50 mg/kg single loading dose of IV levetiracetam

SUMMARY:
The primary objective of this study is to determine the pharmacokinetic profile of a 50 mg/kg loading dose of intravenous levetiracetam (LEV) in term and late preterm infants with seizures. Secondary objectives are to evaluate the safety and efficacy of a 50 mg/kg loading dose of levetiracetam in term and preterm infants with seizures, and to obtain data on steady state drug levels of levetiracetam in neonates.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥ 32 weeks
* Postnatal age ≤ 30 days
* Birth weight ≥ 2000 grams
* Admitted to the Neonatal Intensive Care Unit at Cincinnati Children's Hospital
* Clinical or electrographic seizures of any etiology
* Seizures or seizure prophylaxis requiring treatment with levetiracetam
* Parental consent obtained

Exclusion Criteria:

* Infants with renal insufficiency indicated by serum creatinine > 2.0 at any time
* Infants who have previously received levetiracetam
* Parents refuse consent
* Attending physician does not wish the infant to be enrolled in the study
* Infants who are currently receiving an investigational drug

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Merhar, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from 9/2010 to 8/2011 from the NICU at Cincinnati Children's Hospital.
Groups:
- Single Arm, 50 mg/kg of Levetiracetam: Single arm, 50 mg/kg of levetiracetam
Period: Overall Study
Arm/Group | Single Arm, 50 mg/kg of Levetiracetam
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm, 50 mg/kg of Levetiracetam
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Profile
Description: 3 levels for levetiracetam and its metabolite L057 will be drawn: at 5-20 minutes after the dose, 1-2 hours after the dose, and 6-10 hours after the dose. In infants who remain on maintenance doses of the medication, a steady state level will be drawn 4-7 days after the loading dose. Outcome reported is clearance. The median maximum clearance rate was measured in each participant and determined by evaluating the levels of levetiracetam at each time point using MW Pharm.
Time Frame: 5-20 minutes after the dose, 1-2 hours after the dose, 6-10 hours after the dose, and possibly 4-7 days after loading dose (if infants remained on maintenance doses)
Population: all participants had adequate levels drawn for analysis
Measure: Median (Full Range); unit: ml/min/kg
Arm/Group | Single Arm, 50 mg/kg of Levetiracetam
Number analyzed (Participants) | 7
ml/min/kg | 0.51 (0) [0.42 to 0.62]

ADVERSE EVENTS:
Time Frame: 24 hours after dose
Arm/Group | Single Arm, 50 mg/kg of Levetiracetam
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No